CLINICAL TRIAL: NCT02691806
Title: New Indices for Prediction of Human Fatigue During Training Based on Non-invasive Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-16-2918-HS-CTIL
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Muscle Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- research arm (Experimental): Each of the 14 participants will undergo the same 2 days experimental protocol, separated by at least 2 days rest.
  Interventions: Other: experimental protocol

INTERVENTIONS:
Other: experimental protocol — first day- VO2max test with the following measurements: anaerobic threshold, maximum oxygen consumption, heart rate and breathing indices.
  second day- performing the same physical protocol of VO2max test with the measurements: leg muscles activity using a wireless EMG, hemodynamic measurements of oxygen levels in the skin and skin perfusion, the two latest using optic sensors.

SUMMARY:
Sometimes, during strenuous aerobic activity, activity ceases only when the discomfort that follows lack of oxygen would be intolerable. Reaching this fatigue condition can cause organ damage, muscular damage and / or in different tissues of the body. In this study, investigators aim at developing new indexes, based on hemodynamics measurements from the peripheral micro - circulation system, for the benefit of early detection of fatigue during accelerated physical activity.

DETAILED DESCRIPTION:
14 healthy volunteers, 7 males and 7 females, aged 18-30 will participate in this study.The study includes 2 stages: In the first stage, aerobic capacity of the subjects will be measured by measuring maximum oxygen consumption (VO2max test). This phase will be conducted to determine physical measurements that could indicate different stages in muscle fatigue (anaerobic threshold, maximum oxygen consumption, heart rate and breathing indices).

In the second phase, the subjects will perform the same physical effort protocol that carried out at the first stage. Non- invasive measurements of leg muscles activity during aerobic exercise and at rest (before and after activity), will be carried out using a wireless EMG. Additionally, hemodynamic measurements of oxygen levels in the skin and skin perfusion monitoring before and after strenuous activity will be performed using two optic sensors.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-30 years.
* Healthy civilian volunteers.
* Without known medical illness or medication use that might endanger the participants.

Exclusion Criteria:

* The existence or suspicion of existing cardiac or respiratory disease.
* Any metabolic disorder.
* Any muscles or skeleton condition.
* Any neurological condition.
* the physician decision.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
electric activity of leg muscles | 1 day
  the electric activity of leg muscles will be measured using 4 EMG electrodes, 2 in each leg (muscular twins and quadriceps muscle).

SECONDARY OUTCOMES:
oxygen levels in the skin | 1 day
  oxygen levels in the skin will be measured using optic sensor at each leg in the muscular twins area.
anaerobic threshold | 1 day
  anaerobic threshold value is measured using a metabolic system (ERGOTEST 680, ZAN, GERMANY ) during VO2max test.
maximum oxygen consumption | 1 day
  oxygen consumption (VO2) will be monitored continuously using a metabolic system (ERGOTEST 680, ZAN, GERMANY ) during VO2max test.
heart rate | 2 days
  The heart rate will be monitored using a wearable heart rate monitor (Polar® sensor and heart rate monitor watch).
skin perfusion | 1 day
  skin perfusion (changes in blood volume) will be measured using Laser Doppler flowmetry (LDF) of Perimed system at each leg in the muscular twins area.

CONTACTS AND LOCATIONS:
Overall Officials: Haggai Schermann, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Ramat- Gan, Israel

IPD SHARING:
Plan to Share IPD: No